CLINICAL TRIAL: NCT03884452
Title: A Phase III Efficacy And Safety Study of Ezetimibe (SCH58235) 10 mg in Addition to Atorvastatin or Simvastatin in the Therapy of Homozygous Familial Hypercholesterolemia
Brief Title: Ezetimibe (SCH 58235) Taken With Either Atorvastatin or Simvastatin in Participants With Familial Hypercholesterolemia (MK-0653-018)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P01030; P01030 (Other: Schering-Plough Protocol Number); MK-0653-018 (Other: Merck Protocol Number)
Record Dates: First submitted 2019-03-06; First posted 2019-03-21 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2022-02

CONDITIONS: Familial Hypercholesterolemia
MeSH Terms: conditions — Hyperlipoproteinemia Type II | interventions — Atorvastatin; Simvastatin; Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Atorvastatin 80 mg (Experimental): 80 mg atorvastatin taken orally, once daily for 12 weeks
  Interventions: Drug: Atorvastatin; Drug: Placebo for Ezetimibe
- Ezetimibe + Atorvastatin 40 mg (Experimental): 10 mg ezetimibe and 40 mg atorvastatin taken orally, once daily for 12 weeks
  Interventions: Drug: Atorvastatin; Drug: Ezetimibe
- Ezetimibe + Atorvastatin 80 mg (Experimental): 10 mg ezetimibe and 80 mg atorvastatin taken orally, once daily for 12 weeks
  Interventions: Drug: Atorvastatin; Drug: Ezetimibe
- Simvastatin 80 mg (Experimental): 80 mg simvastatin taken orally, once daily for 12 weeks
  Interventions: Drug: Simvastatin; Drug: Placebo for Ezetimibe
- Ezetimibe + Simvastatin 40 mg (Experimental): 10 mg ezetimibe and 40 mg simvastatin taken orally, once daily for 12 weeks
  Interventions: Drug: Simvastatin; Drug: Ezetimibe
- Ezetimibe + Simvastatin 80 mg (Experimental): 10 mg ezetimibe and 80 mg simvastatin taken orally, once daily for 12 weeks
  Interventions: Drug: Simvastatin; Drug: Ezetimibe

INTERVENTIONS:
Drug: Atorvastatin — Tablets taken orally once daily in the morning
  Arms: Atorvastatin 80 mg; Ezetimibe + Atorvastatin 40 mg; Ezetimibe + Atorvastatin 80 mg
Drug: Simvastatin — Tablets taken orally once daily in the morning or evening
  Arms: Ezetimibe + Simvastatin 40 mg; Ezetimibe + Simvastatin 80 mg; Simvastatin 80 mg
Drug: Ezetimibe — Tablet taken orally once daily in the morning or evening
  Arms: Ezetimibe + Atorvastatin 40 mg; Ezetimibe + Atorvastatin 80 mg; Ezetimibe + Simvastatin 40 mg; Ezetimibe + Simvastatin 80 mg
Drug: Placebo for Ezetimibe — Tablets taken orally once daily in the morning or evening
  Arms: Atorvastatin 80 mg; Simvastatin 80 mg

SUMMARY:
The primary objective of this study is to evaluate the efficacy and the safety of ezetimibe (SCH 58235) co-administered with either atorvastatin or simvastatin in participants with homozygous familial hypercholesterolemia (FH).

ELIGIBILITY:
Inclusion Criteria:

* With a diagnosis of homozygous familial hypercholesterolemia
* All females must have a negative pregnancy test prior to study entry. Women of child bearing potential must agree to practice an effective barrier method of birth control for the duration of the study, until one month after treatment.
* Postmenopausal women who are receiving postmenopausal hormonal therapy or raloxifene must be maintained on a stable estrogen (ERT), estrogen/progestin (HRT) or raloxifene regimen during the study period. ERT, HRT or raloxifene cannot be changed during study period.
* Must follow prescribed or stricter diet, and demonstrate completion of Diet Diaries

Exclusion Criteria:

* A history of mental instability, drug or alcohol abuse; or have been treated or are being treated for severe psychiatric illness which, in the opinion of the Investigator, may interfere with optimal participation in the study.
* With underlying disease likely to limit life span to less than 1 year.
* Have previously been randomized in any studies examining ezetimibe
* Pregnant or lactating women.
* With known hypersensitivity or any contraindication to statin therapy.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2000-05-03 (Actual); Primary Completion 2001-05-24 (Actual); Study Completion 2001-05-24 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline in Low Density Lipoprotein Cholesterol (LDL-C) measured directly | Baseline and Up to Week 12
Percentage of participants with an Adverse Event (AE) | Up to Week 12

SECONDARY OUTCOMES:
Percent change from baseline in calculated LDL-C | Baseline and Up to Week 12
Percent change from baseline in Total Cholesterol (TC) | Baseline and Up to Week 12
Percent change from baseline in Triglycerides (TG) | Baseline and Up to Week 12
Percent change from baseline in High-density-lipoprotein cholesterol (HDL-C) | Baseline and Up to Week 12
Percent change from baseline in High-density-lipoprotein 2 cholesterol (HDL2-C) | Baseline and Up to Week 12
Percent change from baseline in High-density-lipoprotein 3 cholesterol (HDL3-C) | Baseline and Up to Week 12
Percent change from baseline in Apolipoprotein A-I (Apo A-I) | Baseline and Up to Week 12
Percent change from baseline in Apolipoprotein B (Apo B) | Baseline and Up to Week 12
Percent change from baseline in Lipoprotein(a) [Lp(a)] | Baseline and Up to Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gagne C, Gaudet D, Bruckert E; Ezetimibe Study Group. Efficacy and safety of ezetimibe coadministered with atorvastatin or simvastatin in patients with homozygous familial hypercholesterolemia. Circulation. 2002 May 28;105(21):2469-75. doi: 10.1161/01.cir.0000018744.58460.62. PMID 12034651